CLINICAL TRIAL: NCT02851121
Title: Study of Neurophysiological Correlates of the Link Between Perception and Action Through Varied Protocols of Sensorimotor Studies
Brief Title: Study of Neurophysiological Correlates of the Link Between Perception and Action
Acronym: PSM_EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC14.420
Record Dates: First submitted 2016-07-27; First posted 2016-08-01 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteer
Keywords: Neurophysiological; Perception-action; Link
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other)
  Interventions: Other: Sensorial stimulations; Other: Experimental protocols; Behavioral: Emotional protocols; Other: Protocol with a spatial dimension

INTERVENTIONS:
Other: Sensorial stimulations
Other: Experimental protocols
Behavioral: Emotional protocols
Other: Protocol with a spatial dimension

SUMMARY:
The main goal of this study is to better understand the link between motor system (action) and perception in variable sensorial forms by examining the time course and the dynamic of electroencephalography (EEG) activations. To do so, differents sensimotor study protocols in linguistics and in the fiels of emotional and spatial perception will be realised in order to study prcisely differents links parception-action.

ELIGIBILITY:
Inclusion Criteria:

* Signed free consent
* Medical exam done before participation to the study
* Age between 18 and 65 years
* Baccalaureate as minimum degree level

Exclusion Criteria:

* Subject already taking part in an other clinical and/or therapeutic trial still in progress
* Important audition or visual disorder
* Language disorders (aphasia, dysphasia, dysarthria, stammer, etc)
* Any counter-argument to MRI
* Pregnant, parturient or brest feeding women. A pregnancy test (urinary) will be offered to female participants during the inclusion medical interview. In the event of a refusal the woman will have to sign a discharge attesting that she doesn't take any risk of getting pregnant and to volunteer to participate to the trial without having recourse to the offered prgnancy test.
* Patient derpived of liberty by a judicial or administrative decision
* Patient under 18 years under a legal protection or unable to express their consent
* Alcohol ingested

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | 20 minutes
  Software : Brain Analyzer. Hz
Electrooculography (EOG) | Half an hour
  mV
Electromyography EMG | Half an hour
  EMG Delsys sans fil Trigno Digital system. mV
Electrodermal conductance | Half an hour
  EDA device from BrainProduct society. Constant voltage of 0,5V
Anatomical MRI | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Verceuil, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Barsalou LW. Grounded cognition. Annu Rev Psychol. 2008;59:617-45. doi: 10.1146/annurev.psych.59.103006.093639. PMID 17705682
- [Background] Beffara B, Ouellet M, Vermeulen N, Basu A, Morisseau T, Mermillod M. Enhanced embodied response following ambiguous emotional processing. Cogn Process. 2012 Aug;13 Suppl 1:S103-6. doi: 10.1007/s10339-012-0468-6. PMID 22802035
- [Background] Bellier, L., Mazzuca, M., Thai-Van, H., Caclin, A. & Laboissière, R. (2013). Categorization of speech in early auditory evoked responses. INTERSPEECH, page 911-915. ISCA, (2013)
- [Background] Bradley MM, Codispoti M, Cuthbert BN, Lang PJ. Emotion and motivation I: defensive and appetitive reactions in picture processing. Emotion. 2001 Sep;1(3):276-98. PMID 12934687
- [Background] Brandt T, Bartenstein P, Janek A, Dieterich M. Reciprocal inhibitory visual-vestibular interaction. Visual motion stimulation deactivates the parieto-insular vestibular cortex. Brain. 1998 Sep;121 ( Pt 9):1749-58. doi: 10.1093/brain/121.9.1749. PMID 9762962
- [Background] Campagne A, Pebayle T, Muzet A. Oculomotor changes due to road events during prolonged monotonous simulated driving. Biol Psychol. 2005 Mar;68(3):353-68. doi: 10.1016/j.biopsycho.2004.05.003. PMID 15620799
- [Background] Campagne, A., Petit-Boulanger, C., Pebayle, T., Muzet, A., Priez, A. (2004). Electrodermal responses according to mental and emotional loads in driving situations: influence of workload. International Conference on Traffic and Transport Psychology, Nottingham, 5-9 September 2004.
- [Background] Cheetham M, Pedroni AF, Antley A, Slater M, Jancke L. Virtual milgram: empathic concern or personal distress? Evidence from functional MRI and dispositional measures. Front Hum Neurosci. 2009 Oct 20;3:29. doi: 10.3389/neuro.09.029.2009. eCollection 2009. PMID 19876407
- [Background] Collet C, Dittmar A, Vernet-Maury E. Programming or inhibiting action: evidence for differential autonomic nervous system response patterns. Int J Psychophysiol. 1999 Jun;32(3):261-76. doi: 10.1016/s0167-8760(99)00022-7. PMID 10437637
- [Background] D'Ausilio A, Pulvermuller F, Salmas P, Bufalari I, Begliomini C, Fadiga L. The motor somatotopy of speech perception. Curr Biol. 2009 Mar 10;19(5):381-5. doi: 10.1016/j.cub.2009.01.017. Epub 2009 Feb 12. PMID 19217297
- [Background] Decety, J., & Lamm, C. (2009). The biological basis of empathy. In J. T. Cacioppo & Bernston, G. G. (Eds.), Handbook of Neuroscience for the Behavioral Sciences. New York: John Wiley and Sons.
- [Background] Dichgans JM, Brandt T (1978). Visual-vestibular interaction: effect on self-motion and postural control. In R. Held, H. W. Leibowitz, & H. L. Teuber (Eds.), Handbook of Sensory Physiology (Vol. 8, pp. 755-804). Berlin: Springer.
- [Background] Fradcourt B. (2014). Caractérisation du traitement visuel de scènes naturelles émotionnelles : Evaluations comportementales et en Imagerie par Résonance Magnétique fonctionnelle. Thèse de doctorat, Grenoble.
- [Background] Galantucci B, Fowler CA, Turvey MT. The motor theory of speech perception reviewed. Psychon Bull Rev. 2006 Jun;13(3):361-77. doi: 10.3758/bf03193857. PMID 17048719
- [Background] Goubert L, Craig KD, Vervoort T, Morley S, Sullivan MJL, Williams CAC, Cano A, Crombez G. Facing others in pain: the effects of empathy. Pain. 2005 Dec 5;118(3):285-288. doi: 10.1016/j.pain.2005.10.025. Epub 2005 Nov 14. No abstract available. PMID 16289804
- [Background] Goubert L, Eccleston C, Vervoort T, Jordan A, Crombez G. Parental catastrophizing about their child's pain. The parent version of the Pain Catastrophizing Scale (PCS-P): a preliminary validation. Pain. 2006 Aug;123(3):254-263. doi: 10.1016/j.pain.2006.02.035. Epub 2006 Apr 27. PMID 16644128
- [Background] Guenther FH. Cortical interactions underlying the production of speech sounds. J Commun Disord. 2006 Sep-Oct;39(5):350-65. doi: 10.1016/j.jcomdis.2006.06.013. Epub 2006 Aug 2. PMID 16887139
- [Background] Howard I P, Cheung BSK, Landolt J (1987). Influence of vection axis and body posture on visually induced self-rotation and tilt. Advisory Group for Aerospace Research and Development, 433, 15-1-15-8.
- [Background] Jackson PL, Meltzoff AN, Decety J. How do we perceive the pain of others? A window into the neural processes involved in empathy. Neuroimage. 2005 Feb 1;24(3):771-9. doi: 10.1016/j.neuroimage.2004.09.006. PMID 15652312
- [Background] Jackson PL, Rainville P, Decety J. To what extent do we share the pain of others? Insight from the neural bases of pain empathy. Pain. 2006 Nov;125(1-2):5-9. doi: 10.1016/j.pain.2006.09.013. Epub 2006 Sep 25. No abstract available. PMID 16997470
- [Background] Kennedy, R.S., Lane, N.E., Berbaum, K.S., & Lilienthal, M.G. (1993). Simulator Sickness Questionnaire (SSQ): A new method for quantifying simulator sickness. International Journal of Aviation Psychology, 3(3), 203-220.
- [Background] Kleinschmidt A, Thilo KV, Buchel C, Gresty MA, Bronstein AM, Frackowiak RS. Neural correlates of visual-motion perception as object- or self-motion. Neuroimage. 2002 Aug;16(4):873-82. doi: 10.1006/nimg.2002.1181. PMID 12202076
- [Background] Kuhl PK, Conboy BT, Coffey-Corina S, Padden D, Rivera-Gaxiola M, Nelson T. Phonetic learning as a pathway to language: new data and native language magnet theory expanded (NLM-e). Philos Trans R Soc Lond B Biol Sci. 2008 Mar 12;363(1493):979-1000. doi: 10.1098/rstb.2007.2154. PMID 17846016
- [Background] Lamm C, Batson CD, Decety J. The neural substrate of human empathy: effects of perspective-taking and cognitive appraisal. J Cogn Neurosci. 2007 Jan;19(1):42-58. doi: 10.1162/jocn.2007.19.1.42. PMID 17214562
- [Background] Lang PJ, Greenwald MK, Bradley MM, Hamm AO. Looking at pictures: affective, facial, visceral, and behavioral reactions. Psychophysiology. 1993 May;30(3):261-73. doi: 10.1111/j.1469-8986.1993.tb03352.x. PMID 8497555
- [Background] Lavigne KM, Rapin LA, Metzak PD, Whitman JC, Jung K, Dohen M, Loevenbruck H, Woodward TS. Left-dominant temporal-frontal hypercoupling in schizophrenia patients with hallucinations during speech perception. Schizophr Bull. 2015 Jan;41(1):259-67. doi: 10.1093/schbul/sbu004. Epub 2014 Feb 19. PMID 24553150
- [Background] Lotto AJ, Hickok GS, Holt LL. Reflections on mirror neurons and speech perception. Trends Cogn Sci. 2009 Mar;13(3):110-4. doi: 10.1016/j.tics.2008.11.008. Epub 2009 Feb 14. PMID 19223222
- [Background] Mathieu N. (2013). Traitement neurocognitif des émotions au cours du vieillissement: étude de l'"effet de positivité" et ses conséquences. Évaluations comportementales et électroencéphalographiques. Thèse de doctorat
- [Background] Mathieu NG, Gentaz E, Harquel S, Vercueil L, Chauvin A, Bonnet S, Campagne A. Brain processing of emotional scenes in aging: effect of arousal and affective context. PLoS One. 2014 Jun 16;9(6):e99523. doi: 10.1371/journal.pone.0099523. eCollection 2014. PMID 24932857
- [Background] MILGRAM S. BEHAVIORAL STUDY OF OBEDIENCE. J Abnorm Psychol. 1963 Oct;67:371-8. doi: 10.1037/h0040525. No abstract available. PMID 14049516
- [Background] Milgram, S. (1974). Obedience to authority: An experimental view. New York: Harper & Row.
- [Background] Moulin-Frier, C., Laurent, R., Bessière, P., Schwartz, J.L. & Diard, J. (2012). Adverse conditions improve distinguishability of auditory, motor and perceptuo-motor theories of speech perception: an exploratory bayesian modeling study. Lang. Cognitive Proc., 27, 1240-1263.
- [Background] Niedenthal PM. Embodying emotion. Science. 2007 May 18;316(5827):1002-5. doi: 10.1126/science.1136930. PMID 17510358
- [Background] Niedenthal PM, Mermillod M, Maringer M, Hess U. The Simulation of Smiles (SIMS) model: Embodied simulation and the meaning of facial expression. Behav Brain Sci. 2010 Dec;33(6):417-33; discussion 433-80. doi: 10.1017/S0140525X10000865. PMID 21211115
- [Background] Pulvermuller F, Fadiga L. Active perception: sensorimotor circuits as a cortical basis for language. Nat Rev Neurosci. 2010 May;11(5):351-60. doi: 10.1038/nrn2811. Epub 2010 Apr 9. PMID 20383203
- [Background] Rapin LA, Dohen M, Loevenbruck H, Whitman JC, Metzak PD, Woodward TS. Hyperintensity of functional networks involving voice-selective cortical regions during silent thought in schizophrenia. Psychiatry Res. 2012 May 31;202(2):110-7. doi: 10.1016/j.pscychresns.2011.12.014. Epub 2012 Jun 14. PMID 22703623
- [Background] Rapin L, Dohen M, Polosan M, Perrier P, Loevenbruck H. An EMG study of the lip muscles during covert auditory verbal hallucinations in schizophrenia. J Speech Lang Hear Res. 2013 Dec;56(6):S1882-93. doi: 10.1044/1092-4388(2013/12-0210). PMID 24687444
- [Background] Schwartz, J.; Basirat, A.; Ménard, L. & Sato, M. (2012) The Perception-for-Action-Control Theory (PACT): A perceptuo-motor theory of speech perception. Journal of Neurolinguistics, 25, 336-354.
- [Background] Siddle DA, Lipp OV, Dall PJ. The effects of task type and task requirements on the dissociation of skin conductance responses and secondary task probe reaction time. Psychophysiology. 1996 Jan;33(1):73-83. doi: 10.1111/j.1469-8986.1996.tb02110.x. PMID 8570797
- [Background] Singer T, Seymour B, O'Doherty J, Kaube H, Dolan RJ, Frith CD. Empathy for pain involves the affective but not sensory components of pain. Science. 2004 Feb 20;303(5661):1157-62. doi: 10.1126/science.1093535. PMID 14976305
- [Background] Skipper JI, van Wassenhove V, Nusbaum HC, Small SL. Hearing lips and seeing voices: how cortical areas supporting speech production mediate audiovisual speech perception. Cereb Cortex. 2007 Oct;17(10):2387-99. doi: 10.1093/cercor/bhl147. Epub 2007 Jan 11. PMID 17218482
- [Background] Stern JA, Boyer D, Schroeder D. Blink rate: a possible measure of fatigue. Hum Factors. 1994 Jun;36(2):285-97. doi: 10.1177/001872089403600209. PMID 8070793
- [Background] Tanahashi S, Ujike H, Ukai K. Visual rotation axis and body position relative to the gravitational direction: Effects on circular vection. Iperception. 2012;3(10):804-19. doi: 10.1068/i0479. Epub 2012 Dec 4. PMID 23483823
- [Background] Vermeulen N, Pleyers G, Mermillod M. Second-person social neuroscience: connections to past and future theories, methods, and findings. Behav Brain Sci. 2013 Aug;36(4):440-1. doi: 10.1017/S0140525X12002075. PMID 23883770
- [Background] Vermeulen N, Chang B, Corneille O, Pleyers G, Mermillod M. Verifying properties of concepts spontaneously requires sharing resources with same-modality percept. Cogn Process. 2013 Mar;14(1):81-7. doi: 10.1007/s10339-012-0533-1. Epub 2013 Feb 15. PMID 23413000